CLINICAL TRIAL: NCT00725335
Title: The Effect of Ischemia/Reperfusion Injuries Elicited by Pringle Manoeuvre on the Prognosis of HCC Patients After Curative Excision:A Multicenter Prospective Randomized Controlled Trial
Brief Title: Effect of I/R Injuries by Pringle Manoeuvre on the Prognosis of HCC Patients After Curative Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Collaborators: Chinese PLA General Hospital (Other); Fudan University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, feng xiaobin, Dr Feng xiaobin, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWHB001; ISRCTN01960869 (Other: a organization in UK)
Record Dates: First submitted 2008-07-24; First posted 2008-07-30 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: ischemia; liver cancer; radical excision; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Ischemia; Liver Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A,non-pringle group (Experimental): Intervention of curative resection of HCC Without pringle manoeuvre in this arm
  Interventions: Procedure: curative resection without Pringle
- pringle group(B) (Active Comparator): when the curative resection of HCC performed, the pringle manoeuvre will be routinely applied.
  Interventions: Procedure: curative resection with Pringle manoeuvre

INTERVENTIONS:
Procedure: curative resection without Pringle — Radical excision of liver cancer without the procedure of pringle manoeuvre
  Other Names: Experimental group
  Arms: group A,non-pringle group
Procedure: curative resection with Pringle manoeuvre — curative resection liver cancer under pringle manoeuvre
  Other Names: control group
  Arms: pringle group(B)

SUMMARY:
This is a multi-centre prospective randomized controlled trial to explore the influence of ischemia-reperfusion injuries elicited by pringle manoeuvre during radical excision on the prognosis of Hepatocellular Carcinoma (HCC) patients.

DETAILED DESCRIPTION:
Until now there are two popular procedures during the radical excision of primary liver cancer in our country.One is to give a pringle manoeuvre to control the operative blood loss,the other is using a combination of CUSA and Tissue-link to control the bleeding while without liver ischemia.According to the recent experimental studies in rats,we know that the ischemia and reperfusion injury may contribute to the metastasis of the tumor.In order to test the actual contribution of ischemia on human,we conduct this prospective clinical trial to compare the two popular procedures' effect on the prognosis of liver cancer patients undergoing radical excision.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of resectable primary liver cancer
* The liver function showed:Child-Pugh A，ICG-R15 < 20%
* HbsAg (+)
* tumor nodes in the liver were singular or multiple and could be radical excision
* No preoperative anti-cancer therapy
* Written informed consent from the patient or legal guardian prior to entering the study

Exclusion Criteria:

* Pregnancy patients
* With extrahepatic tumor or lymphnode metastasis
* Tumor invasion or thrombosis in portal vein,hepatic vein or inferior vena cava
* Positive marginal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 1,3,5-year

SECONDARY OUTCOMES:
overall survival,morbidity,postoperative mortality;blood loss,Liver function test,etc | baseline~2 weeks, 5-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jiahong, Ph D, Study Director — Institue of hepatobiliary surgery,Chinese PLA General Hospital
Locations (1):
- Institute of hepatobiliary surgery,southwest hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Xiaobin F, Shuguo Z, Jian Z, Yudong Q, Lijian L, Kuansheng M, Xiaowu L, Feng X, Dong Y, Shuguang W, Ping B, Jiahong D. Effect of the pringle maneuver on tumor recurrence of hepatocellular carcinoma after curative resection (EPTRH): a randomized, prospective, controlled multicenter trial. BMC Cancer. 2012 Aug 3;12:340. doi: 10.1186/1471-2407-12-340. PMID 22862951
- See also: Protocol — http://www.ncbi.nlm.nih.gov/pubmed/22862951